CLINICAL TRIAL: NCT05918640
Title: Lurbinectedin in FET-Fusion Tumors (LIFFT)
Brief Title: Lurbinectedin in FET-Fused Tumors
Acronym: LiFFT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Jazz Pharmaceuticals (Industry); Stand Up To Cancer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-020814
Record Dates: First submitted 2023-06-06; First posted 2023-06-26 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Ewing Sarcoma; Desmoplastic Small Round Cell Tumor; Pediatric Cancer; Undifferentiated Sarcoma
Keywords: Ewing Sarcoma-Friend Leukemia Integration 1 Transcription factor (ESW-FLI1); Ewing Sarcoma Breakpoint Region 1-Friend Leukemia Integration 1 Transcription factor (EWSR1-FLI1); Ewing Sarcoma Erythroblast Transformation Specific Related Gene (EWS-ERG); Ewing Sarcoma Breakpoint Region 1 (EWRS1); TATA-Box-Binding Protein Associated Factor 15 (TAF15); Fused Tumors (FET); Ewing Sarcoma-Wilms' Tumor Gene 1 (EWS-WT1)
MeSH Terms: conditions — Sarcoma, Ewing; Desmoplastic Small Round Cell Tumor; Neoplasms | interventions — PM 01183

STUDY DESIGN:
Intervention Model Description: The first part of this study is a standard 3+3 design to test the safety, tolerability and pharmacokinetic profile of lurbinectedin administered on a day 1, 4 schedule in patients with FET-fusion tumors. The second part of this study is a single-stage phase 2 design and will accrue 17 patients in parallel to the exploratory cohort after the Recommended Phase 2 Dose (RP2D) is determined.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ewing Sarcoma (Experimental): The first part of this study is a standard 3+3 design to test the safety, tolerability and pharmacokinetic profile of lurbinectedin administered on a day 1, 4 schedule in patients with FET-fusion tumors.
  Interventions: Drug: Lurbinectedin

INTERVENTIONS:
Drug: Lurbinectedin — Lurbinectedin will be administered on a Day 1, Day 4 schedule every 21 days. Doses will be determined in the phase 1 portion of the trial.

SUMMARY:
The purpose of this study is to find out if a drug called lurbinectedin (the "study drug") is safe and effective at treating people with recurrent or relapsed solid tumors, including Ewing sarcoma.

DETAILED DESCRIPTION:
In this study, the investigators will test the activity of lurbinectedin as a targeted therapy for FET (FUS, Ewing Sarcoma Breakpoint Region 1 (EWRS1), TATA-Box-Binding Protein Associated Factor 15 (TAF15)). Ewing sarcoma is driven by the Ewing Sarcoma-Friend Leukemia Integration 1 Transcription Factor (EWS-FLI1). Lurbinectedin has been shown to inhibit EWS-FLI1 and Ewing Sarcoma-Wilms' Tumor Gene 1 (EWS-WT1) in preclinical models. Therefore, the goal of this study is to see if Lurbinectedin can be used to inhibit EWS-FLI1, EWS-WT1, or other FET fusion proteins to drive tumor responses in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 10 years.
2. Phase 1: Histological confirmed diagnosis of recurrent or relapsed solid tumor failing primary therapy. Patients must have a known FET fusion (fusion that contains EWSR1, FUS, or TAF15) as documented by next generation sequencing, polymerase chain reaction (PCR) or Fluorescence in situ hybridization (FISH). Patients with a histological diagnosis of Ewing sarcoma with EWS-FLI1 are eligible for dose escalation but not for the exploratory cohort. Please note patients with Ewing sarcoma and alternative FET-ETS fusions (including but not limited to EWS-ERG, EWS-ETV1, EWS-ETV4, EWS-FEV, FUS-ERG, FUS-FEV) are eligible for the exploratory cohort.
3. Phase 2: Histologically confirmed diagnosis of recurrent or relapsed Ewing sarcoma failing primary therapy with confirmation of EWS-FLI1 fusion and breakpoint by Next generation sequencing or PCR or EWSR1 rearrangement confirmed by FISH and available tissue for central confirmation of EWS-FLI1 fusion and breakpoint.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2 (age ≥16 years) or Lansky of at least 60 (age <16 years).
5. Disease status (baseline imaging must be performed within 28 days of Day 1 of study treatment):

   1. Phase 1: At least one site of measurable disease on CT or MRI as defined by RECIST 1.1 OR evaluable disease with at least one site of disease that has not been previously radiated
   2. Phase 2: At least one site of measurable disease on CT or MRI as defined by RECIST 1.1
6. Meets organ function requirements as outlined below:

   1. Liver:

      Alanine aminotransferase (ALT) ≤ 2.5X upper limit of normal. For the purposes of this study the upper limit of normal for ALT is 45 U/L. Aspartate aminotransferase (AST) ≤ 2.5X upper limit of normal. For the purposes of this study the upper limit of normal for AST is 50 U/L. Total bilirubin ≤ 1.5X institutional upper limit of normal with the exception of patients with Gilbert's syndrome who must have bilirubin <3X institutional upper limit of normal.
   2. Renal:

      Creatinine Calculated creatinine clearance (by the Schwartz equation for patients <18 years of age and Cockroft-Gault formula (Appendix B) for patients ≥18 years of age) or radionuclide glomerular filtration rate (GFR) ≥ 50 mL/min /m2 or a serum creatinine less than or equal to the age/gender valued below:

      Age Maximum Serum Creatinine (mg/dL) Male Female 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4

      ≥ 16 years 1.7 1.4
   3. Bone marrow:

      Absolute Neutrophil Count (ANC) ≥ 1,000/µL (>one week since last dose of short acting medications (e.g. filgrastim) and > two weeks since last dose of long acting medications (e.g. peg-filgrastim)) Platelet Count (PLTs) ≥ 100,000/ µL (>two weeks since last dose of thrombopoietin receptor agonist such as romiplostim and without platelet transfusion within previous 7 days of screening laboratories) Patients with a history of bone marrow involvement are required to have bilateral bone marrow aspirates and biopsies at baseline. Subjects with bone marrow disease are eligible as long as they meet the hematologic requirements above and are not known to be refractory to red cell or platelet transfusions.
   4. Cardiac:

   Creatine phosphokinase ≤ 2.5 x institutional upper limit of normal, Left ventricular ejection fraction (LVEF) or shortening fraction (SF) per institutional norm LVEF > 50% OR SF >28%.
7. Written, voluntary informed consent
8. Fertile males and females of childbearing potential must agree to use an effective method of birth control from screening, through 6 months after last study drug administration for females and 4 months for males. Women of childbearing potential must have a negative pregnancy test during screening procedures. Effective methods of birth control include: double barrier method (condom, diaphragm), abstinence, an intrauterine device (IUD), levonorgestrol implants, medroxyprogesterone acetate injections, or oral contraception. For those subjects whose preferred and usual lifestyle employs abstinence, refraining from heterosexual intercourse must be practiced during the entire active phase of the trial.
9. Patients ≥18 years must be willing to undergo tumor biopsy at study entry. Patients with Ewing sarcoma or DSRCT must be willing to undergo biopsy post-treatment. If biopsy is contraindicated, enrollment must be approved by study PI and archival tissue must be available.
10. Time elapsed from previous therapy:

    1. Must be ≥ 3 weeks for systemic myelosuppressive therapy
    2. ≥ 2 weeks for local radiation therapy (small field), ≥ 150 days after thyrotropin binding inhibition (TBI), craniospinal external beam radiotherapy (XRT) or radiation to ≥50% of the pelvis
    3. ≥ 2 weeks for major surgery
    4. ≥ 2 weeks for monoclonal antibodies and oral kinase inhibitors.
    5. ≥ 6 weeks for autologous stem cell transplant. 6 months for allogeneic stem cell transplant.
    6. ≥ 6 weeks for any type of cellular therapy
11. Patients must be recovered to baseline or Grade ≤1from the acute adverse effects of prior treatments, with the exception of alopecia and decreased deep tendon reflexes.

Exclusion Criteria:

1. Prior therapy with trabectedin or lurbinectedin.
2. Subjects with known brain metastases.
3. Subjects with a known bleeding diathesis.
4. Subjects who are pregnant or breastfeeding.
5. Concurrent therapy:

   1. Patients who are currently receiving an investigational drug or another anticancer agent
   2. Patients receiving over the counter or herbal supplement with significant potential hepatotoxicity in the opinion of the investigator.
   3. Patients receiving a medically necessary strong or moderate CYP3A4 inhibitor or inducer within 14 days prior to the first dose of study drug.
6. Clinically significant, unrelated illness or uncontrolled infection which would, in the opinion of the treating physician, compromise the patient's ability to tolerate the investigational agents or be likely to interfere with the study procedures or results.
7. Subjects who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study, or in whom compliance is likely to be suboptimal, should be excluded.
8. Patients with known active viral hepatitis (i.e. Hepatitis A, B, or C)

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Dose Limiting Toxicities (DLTs) | within 28 days of the first dose
  First cycle (approximately 21 days) Dose Limiting Toxicities (DLTs) will be evaluated.
Phase 1: Frequency of adverse events | 28 days after last dose
  Adverse events to be reported during treatment and for at least 28 days after last dose.
Phase 1: Complete Response or Partial Response | through the end of treatment, an average of 1 year
  Percentage of participants with complete response or partial response will be assessed approximately every 2 to 4 cycles through the end of treatment and up to at least 28 days after the last dose.
Phase 2: Event-Free Survival (EFS) | 2 years
  Event-free survival (EFS) is based on investigator assessment from baseline until Month 24.

SECONDARY OUTCOMES:
Phase 1: Maximum observed Plasma Concentration (Cmax) | at the end of cycle 1 (each cycle is 28 days)
  Maximum observed plasma concentration (Cmax) will be used to assess Lurbinectedin Pharmacokinetics
Phase 1: Area under the concentration-time curve (AUC) | at the end of cycle 1 (each cycle is 28 days)
  Area under the concentration-time curve (AUC) will be used to assess Lurbinectedin Pharmacokinetics
Phase 2: 6-month Progression Free Survival (PFS) | 6 months
  Progression Free Survival (PFS) assessed from the first dose of study drug to earliest date of death or progressive disease.
Phase 1: Duration of Response (DoR) | Up to 5 years
  Duration of Response (DoR) defined as time from date of first response (Complete Response or Partial Response) in responders to date of progression or death
Phase 2: Overall Survival | Up to 5 years
  Overall survival (OS) defined as the time from enrollment to date of death due to any cause.
Phase 2: Disease Control Rate | Up to 5 Years
  Disease Control ate is defined as the percentage of patients who sustain a complete response, partial response, or stable disease over 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Laetsch, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (6):
- United States (6):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No